CLINICAL TRIAL: NCT07111767
Title: Effectiveness of a Modified Cost-Effective Dietary Plan in Promoting Weight Loss and Preservation of Lean Body Mass in Patients After Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Dr Safina Tanveer, PRINCIPAL INVESTIGATOR| Trainee Medical Officer, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 661/DME/KMC
Record Dates: First submitted 2025-07-28; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Bariatric Surgery; Nutritional Status; Body Composition
Keywords: Bariatric surgery; Obesity management; Post-bariatric diet; Cost-effective diet; Low-cost diet plan; Vitamin B12 deficiency; Iron deficiency; Vitamin D deficiency; Weight loss after bariatric surgery; Lean body mass preservation
MeSH Terms: conditions — Obesity; Vitamin B 12 Deficiency; Iron Deficiencies; Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: Cost-effective Post-Operative diet (Experimental): Participants in this arm will follow a low-cost dietary plan designed according to the American Society for Metabolic and Bariatric Surgery (ASMBS) guidelines, using locally available, affordable foods to meet protein and micronutrient needs. The plan aims to promote weight loss, preserve lean body mass, and prevent nutrient deficiencies.
  Interventions: Dietary Supplement: Low-Cost Post-Bariatric Diet
- Control - Standard High-Cost Postoperative Diet (Active Comparator): Participants in this arm will follow the standard postoperative hospital diet, which includes expensive protein supplements (e.g., whey protein, cottage cheese) and imported nutritional products typically recommended after bariatric surgery.
  Interventions: Dietary Supplement: Standard High-cost Post-Bariatric Diet

INTERVENTIONS:
Dietary Supplement: Low-Cost Post-Bariatric Diet — Low-Cost Post-Bariatric Diet (Experimental):
  Based on the American Society for Metabolic and Bariatric Surgery (ASMBS) guidelines.
  Uses affordable, locally available foods (e.g., eggs, lentils, local dairy products) to meet protein and micronutrient needs.
  Designed to be cost-effective and accessible for patients from low-income or rural areas.
  Arms: Experimental Arm: Cost-effective Post-Operative diet
Dietary Supplement: Standard High-cost Post-Bariatric Diet — Standard Post-Bariatric Diet (Active Comparator):
  The conventional high-cost diet currently followed at the study hospital. Includes imported or expensive protein supplements such as whey protein and cottage cheese, along with nutritional products not easily accessible in rural or low-resource settings.
  Arms: Control - Standard High-Cost Postoperative Diet

SUMMARY:
This study will see if a low-cost dietary plan, based on the standard dietary guidelines of the American Society for Metabolic and Bariatric Surgery (ASMBS) and using locally available foods, can help patients lose weight and keep their lean body mass after bariatric surgery. It will also check if this plan can maintain healthy levels of important nutrients such as vitamin B12, iron, and vitamin D.

Patients who have undergone bariatric surgery will be randomly assigned to follow either the low-cost diet or the regular hospital diet. Their weight, body composition, and nutrient levels will be tracked at baseline, and at 1, 3, and 6 months after surgery.

The aim is to find out if this simpler, affordable diet, which follows international standards, works as well as the regular plan while being easier for low-income patients to follow.

DETAILED DESCRIPTION:
Obesity is a growing global health problem and is recognized by the World Health Organization (WHO) as a leading cause of preventable disease. It is a complex, long-term condition influenced by multiple factors, and treatment options range from lifestyle changes to medications and surgery. Bariatric surgery is currently the most effective long-term treatment for morbid obesity. It not only helps in significant weight loss but also improves obesity-related health problems such as type II diabetes, hypertension, and obstructive sleep apnea, while improving quality of life.

Among the various surgical techniques, Roux-en-Y gastric bypass (RYGB), sleeve gastrectomy (SG), and one-anastomosis gastric bypass (OAGB/MGB) are the most commonly performed. However, these surgeries can lead to reduced absorption of essential nutrients because they bypass parts of the intestine where vitamins and minerals are absorbed. Nutrient deficiencies, particularly in vitamin B12, iron, and vitamin D, are common after bariatric surgery. Therefore, structured dietary management and supplementation are essential after surgery to prevent these deficiencies and preserve lean body mass (LBM).

Standard dietary recommendations from the American Society for Metabolic and Bariatric Surgery (ASMBS) suggest a gradual progression from liquids to solid foods, adequate protein intake (1.0-1.5 g/kg), and lifelong use of vitamin and mineral supplements. However, in countries like Pakistan, where 45% of the population lives below the international poverty line, the standard postoperative diet often includes costly imported supplements like whey protein, which are unaffordable and hard to access for most patients, particularly those from rural areas. This creates barriers to dietary compliance and worsens clinical outcomes.

Adequate protein intake plays a key role in preserving lean body mass and improving recovery after bariatric surgery. Nutritional deficiencies, particularly in vitamin B12, iron, and vitamin D, remain prevalent after bariatric surgery and require targeted nutritional strategies.

In response to these challenges, this study introduces a low-cost dietary plan based on ASMBS guidelines using locally available, affordable foods to meet protein and micronutrient needs. It aims to compare this plan with the conventional high-cost hospital diet to determine whether it can effectively promote weight loss, maintain lean body mass, and prevent micronutrient deficiencies. By aligning with international standards while addressing local socioeconomic constraints, this approach could improve patient adherence, nutritional outcomes, and overall recovery following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed written consent
* Adults between the ages of 18 and 65 undergoing primary bariatric surgery (Roux-en-Y gastric bypass, sleeve gastrectomy, or OAGB)

Exclusion Criteria:

* Patients having revision bariatric surgery
* Patients with recognized diseases related to micronutrient supplementation
* Patients with pre-existing gastrointestinal, metabolic, or endocrine disorders that impair nutrient absorption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | Baseline, 1 month, 3 months, and 6 months after surgery.
  Weight loss will be measured using a calibrated digital weighing scale.Weight loss will be defined as the reduction in body weight (kg) from baseline.
  Unit of Measure: Kilograms (kg)

SECONDARY OUTCOMES:
Change in Serum Iron Levels | Baseline, 1 month, 3 months, and 6 months post-surgery.
  Hemoglobin (g/dL) and serum ferritin (ng/mL) measured via blood tests.Iron deficiency will be defined as Hb <12 g/dL (women) or <13 g/dL (men) and/or ferritin <15 ng/mL.
Change in Serum Vitamin B12 Levels | Baseline, 1 month, 3 months, and 6 months post-surgery.
  Measured via serum vitamin B12 assay.Levels below 200 pg/mL will be considered deficient.
Change in Serum Vitamin D Levels | Baseline, 1 months, 3 months, and 6 months post-surgery.
  Serum 25(OH) vitamin D (ng/mL) measured via blood assay . Levels below 20 ng/mL will be considered deficient.
Lean Body Mass (LBM) | Baseline, 1 month, 3 months, and 6 months postoperatively
  Change in lean body mass assessed using bioelectrical impedance analysis to evaluate preservation of lean tissue after bariatric surgery. Unit of Measure: Kilograms (kg)
Body Mass Index (BMI) | Baseline, 1 month, 3 months, and 6 months postoperatively
  BMI will be calculated by dividing weight (kg) by height squared (m²). Height will be measured only at baseline, as it remains unchanged postoperatively. Follow-up BMI will be derived using baseline height and follow-up weight measurements.Unit of Measure: kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Safina Tanveer, MBBS, FCPS-II, Principal Investigator — Khyber Teaching Hospital
Locations (1):
- Khyber Teaching Hospital, Peshawar, Khyber Pakhtun Khwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Via MA, Mechanick JI. Nutritional and Micronutrient Care of Bariatric Surgery Patients: Current Evidence Update. Curr Obes Rep. 2017 Sep;6(3):286-296. doi: 10.1007/s13679-017-0271-x. PMID 28718091
- See also: Evidence-based guidelines from ASMBS on nutritional and micronutrient management for bariatric surgery patients, including dietary progression, protein intake, and supplementation strategies. — https://pubmed.ncbi.nlm.nih.gov/28718091/